CLINICAL TRIAL: NCT00313820
Title: A 13-Week, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel-Group Study To Evaluate The Efficacy, Safety And Tolerability Of Pregabalin (150-600 Mg/Day) Using A Flexible Dosing Schedule In The Treatment Of Subjects With Central Post-Stroke Pain (CPSP)
Brief Title: Efficacy Of Pregabalin In Subjects With Post-Stroke Central Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081063
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2009-10-09 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2009-10

CONDITIONS: Central Neuropathic Pain
Keywords: Post-stroke pain, pregabalin
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): The change from in pain scores from baseline to endpoint among stroke subjects receiving pregabalin will be compared to change in pain scores from baseline to endpoint among stroke subjects receiving matched placebo.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): The change in pain scores from baseline to endpoint will be compared among the two treatment groups- ie subjects receiving 12 weeks of pregabalin treatment vs subjects receiving 12 weeks of placebo treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Eligible subjects with post-stroke central pain will be randomized to receive double blinded treatment using pregabalin or matched placebo. The effects of pregabalin as compared to placebo on pain pain symptoms will be compared over the 13 week clinical trial. At baseline following pain ratings and clinical measures, subjects randomized to pregabalin receive instructions to take 75mg twice a day for 7days. The dosing of pregabalin or matching placebo will be titrated over the first 4 weeks (based on tolerability and pain scores). (Range 150-600mg) After the 4th week, the dose of medication will be maintained until week 12 (when tapering of medication begins) Ratings of Pain severity, review of pain/sleep diaries as well as medication tolerance occur bi-weekly throughout the study. Tapering off med occurs from week 12-13.
  Arms: Pregabalin
Drug: Placebo — Eligible subjects with post-stroke central pain will be randomized to receive double blinded treatment using pregabalin or matched placebo. The effects of pregabalin as compared to placebo on pain pain symptoms will be compared over the 13 week clinical trial. At baseline following pain ratings and clinical measures, subjects randomized to pregabalin receive instructions to take 75mg twice a day for 7days. The dosing of pregabalin or matching placebo will be titrated over the first 4 weeks (based on tolerability and pain scores). (Range 150-600mg) After the 4th week, the dose of medication will be maintained until week 12 (when tapering of medication begins) Ratings of Pain severity, review of pain/sleep diaries as well as medication tolerance occur bi-weekly throughout the study. Tapering off med occurs from week 12-13.
  Arms: Placebo

SUMMARY:
Efficacy and Safety of flexibly dosed pregabalin compared to placebo among subjects with central post stroke pain (CPSP)

ELIGIBILITY:
Inclusion Criteria:

* Positive history of clinical stroke at least 4 months prior to randomization CPSP--3 months prior to screening

Exclusion Criteria:

* History of dementia or any other severe cognitive impairment
* Diabetic Peripheral Neuropathy (DPN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Australia (7):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, East Gosford, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Warrawong, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Footscray, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- China (3):
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Shanghai
- Pfizer Investigational Site, New Territories, Hong Kong
- India (4):
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, Chennai
  - Pfizer Investigational Site, Lucknow
  - Pfizer Investigational Site, New Delhi
- Indonesia (2):
  - Pfizer Investigational Site, Jakarta
  - Pfizer Investigational Site, Surabaya
- Malaysia (3):
  - Pfizer Investigational Site, George Town
  - Pfizer Investigational Site, Kuala Lumpur
  - Pfizer Investigational Site, Kuala Selangor
- Pakistan (2):
  - Pfizer Investigational Site, Karachi, Sindh
  - Pfizer Investigational Site, Karachi
- Pfizer Investigational Site, Manila, Philippines
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (3):
  - Pfizer Investigational Site, Gueishan Shiang, Taoyuan Hsien
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Ratchatewee, Bangkok
  - Pfizer Investigational Site, Bangkok

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081063&StudyName=Efficacy%20Of%20Pregabalin%20In%20Subjects%20With%20Post-Stroke%20Central%20Neuropathic%20Pain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-week screening and washout phase prior to randomization.
Groups:
- Pregabalin: 75 milligram (mg) capsule by mouth (PO) twice a day (BID) for 7 days. Pregabalin was titrated over the first 4 weeks based on tolerability and pain scores. Range was 150 mg total daily dose to a maximum of 600 mg total daily dose. Week 1: 150 mg BID for 7 days; Weeks 2 through 4: maintained at previous dose level or dose increased or reduced based on tolerability and pain scores (150 mg or 300 mg or 600 mg total daily dose). After the fourth week, dose was maintained until week 12 when dose was tapered to 75 mg BID.
- Placebo: 75 milligram (mg) capsule PO BID for 7 days. Placebo was titrated over the first 4 weeks based on tolerability and pain scores. Range was 150 mg total daily dose to a maximum of 600 mg total daily dose. Week 1: 150 mg BID for 7 days; Weeks 2 through 4: maintained at previous dose level or dose increased or reduced based on tolerability and pain scores (150 mg or 300 mg or 600 mg total daily dose). After the fourth week, dose was maintained until week 12 when dose was tapered to 75 mg BID.
Period: Assigned to Treatment
Arm/Group | Pregabalin | Placebo
Started | 111 | 109
Completed | 110 | 109
Not Completed | 1 | 0
Not completed — Other | 1 | 0
Period: Pregabalin or Placebo Treatment Period
Arm/Group | Pregabalin | Placebo
Started | 110 | 109
Completed | 93 | 90
Not Completed | 17 | 19
Not completed — Adverse Event | 9 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 7
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.8) | 57.1 (10.2) | 58.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 67 | 70 | 137

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score at Endpoint as Measured by Daily Pain Rating Scale (DPRS)
Description: Mean pain score obtained from last 7 available DPRS scores up to and including day of Week 12 visit or early termination (ET) equivalent. DPRS: subject rated 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain. Self-assessment performed daily on awakening prior to taking study medication.
Time Frame: Up to Week 12
Population: Intent to Treat (ITT): received at least 1 dose study medication and completed at least 1 post-baseline assessment. Endpoint = Week 12 or ET
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 108 | 108
scores on scale | 4.8 (0.21) | 5.0 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results: Endpoint Mean Pain Score Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.578, ANCOVA; ANCOVA with treatment and country as factors and baseline pain score as covariate; Mean Difference (Final Values) = -0.2, 95% CI [-0.7 to 0.4], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Modelled Results: Treatment by country interaction; Test type: Superiority or Other; p = 0.294, ANCOVA — Interaction p-value based on adding interaction term to the main model

2. Secondary Outcome: Pain Score as Measured by DPRS
Description: Weekly mean pain score measured by DPRS: subject rated 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain. Self-assessment performed daily on awakening prior to taking study medication.
Time Frame: Week 1, Week 2, Week 3, Week 6, Week 9, and Week 12
Population: ITT; (n) = number of participants with analyzable data at observation for pregabalin and placebo, respectively; weeks as specified in timeframe through Week 12 [ET]
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 109
scores on scale
  Week 1 (n=108, 108) | 5.6 (0.18) | 6.0 (0.18)
  Week 2 (n=104, 106) | 5.3 (0.18) | 5.8 (0.18)
  Week 3 (n=102, 105) | 5.1 (0.18) | 5.6 (0.18)
  Week 6 (n=97, 102) | 4.9 (0.18) | 5.4 (0.18)
  Week 9 (n=98, 97) | 4.8 (0.18) | 5.2 (0.18)
  Week 12 [ET] (n=92, 92) | 4.7 (0.18) | 4.9 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1 Modelled Results; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis — Estimated from a repeated measures linear mixed model with treatment, week, country and treatment by week interaction as factors and baseline value as a covariate. A compound symmetry covariance structure is specified; Mean Difference (Final Values) = -0.3, 95% CI [-0.8 to 0.1], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2 Modelled Results; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-1.0 to 0.0], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3 Modelled Results; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI [-1.1 to -0.1], Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 6 Modelled Results; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI [-1.1 to -0.1], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 9 Modelled Results; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.9 to 0.1], Standard Error of Mean 0.25
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 12 Modelled Results; Test type: Superiority or Other; p = 0.592, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI [-0.6 to 0.4], Standard Error of Mean 0.25

3. Secondary Outcome: Number of Subjects With at Least a 30% Reduction From Baseline in Mean Pain Score at Endpoint
Description: 30% Responder Yes = number of subjects with 30% reduction in mean pain score from baseline to observation; 30% reduction calculated as [(T minus B) divided by B multiplied by 100] < = negative 30. T = endpoint mean pain score (obtained from last 7 available scores from DPRS); B = baseline mean pain score (obtained from average of last 7 daily scores from DPRS). 30% Responder No indicates number of subjects that did not reach 30% reduction in mean pain score.
Time Frame: Baseline, Week 12
Population: ITT; endpoint = Week 12 or ET
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 108 | 108
participants
  30% Responders Yes | 48 | 35
  30% Responders No | 60 | 73
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; 30% Responders; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test comparing pregabalin to placebo adjusted for country under the null hypothesis of no treatment difference

4. Secondary Outcome: Number of Subjects With at Least a 50% Reduction From Baseline in Mean Pain Score at Endpoint
Description: 50% Responder Yes = number of subjects with 50% reduction in mean pain score from baseline to observation; 50% reduction calculated as [(T minus B) divided by B multiplied by 100] < = negative 50. T = endpoint mean pain score (obtained from last 7 available scores from DPRS); B = baseline mean pain score (obtained from average of last 7 daily scores from DPRS). 50% Responder No indicates number of subjects that did not reach 50% reduction in mean pain score.
Time Frame: Baseline, Week 12
Population: ITT; endpoint = Week 12 or ET
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 108 | 108
participants
  50 % Responders Yes | 26 | 22
  50 % Responders No | 82 | 86
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; 50% Responders; Test type: Superiority or Other; p = 0.622, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Weekly Mean Sleep Interference Score From Daily Sleep Diary (Daily Sleep Interference Scale [DSIS])
Description: DSIS: subject rated 11-point numeric scale ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep) during past 24-hour period. Higher score indicates a greater level of sleep disturbance. Self-assessment performed daily on awakening prior to taking study medication. Endpoint calculated as mean of last 7 available scores.
Time Frame: Week 1, Week 2, Week 3, Week 6, Week 9, and Week 12
Population: ITT; (n) = number of subjects with analyzable data at observation for pregabalin and placebo, respectively; endpoint = Week 12 or ET.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 109
scores on scale
  Week 1 (n=108, 108) | 3.6 (0.17) | 4.2 (0.17)
  Week 2 (n=104, 106) | 3.5 (0.17) | 4.0 (0.17)
  Week 3 (n=102, 105) | 3.2 (0.17) | 3.9 (0.17)
  Week 6 (n=98, 102) | 3.0 (0.17) | 3.7 (0.17)
  Week 9 (n=98, 97) | 3.0 (0.17) | 3.4 (0.17)
  Week 12 (n=92, 92) | 3.1 (0.18) | 3.2 (0.18)
  Endpoint [Week 12 or ET] (n=108, 108) | 3.0 (0.19) | 3.1 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Modelled Results; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-1.0 to -0.1], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Modelled Results; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-1.0 to -0.0], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Modelled Results; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-1.2 to -0.2], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 6; Modelled Results; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-1.1 to -0.2], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 9; Modelled Results; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.9 to 0.0], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 12; Modelled Results; Test type: Superiority or Other; p = 0.663, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI [-0.6 to 0.4], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Endpoint [Week 12 or ET]; Modelled Results; Test type: Superiority or Other; p = 0.627, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI [-0.6 to 0.4], Standard Error of Mean 0.26

6. Secondary Outcome: Short Form-McGill Pain Questionnaire (SF-MPQ Visual Analog Scale [VAS]) - Part B Only
Description: SF-MPQ Part B VAS consists of a line 0 to 100 millimeters (mm) in length; range is (no pain) to 100 mm (worst possible pain). Subjects placed a mark indicating the intensity of their pain. Distance from left-hand end of line was measured and entered on Case Report Form (CRF) as score in mm. Higher score indicates greater level of pain.
Time Frame: Week 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 97
millimeters | 48.5 (2.19) | 49.5 (2.23)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.741, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline value as a covariate; Mean Difference (Final Values) = -1.0, 95% CI [-7.0 to 5.0], Standard Error of Mean 3.05

7. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI: subject rated questionnaire to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]). Includes 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each of the relevant dimensions and a total score (0 to 100). Higher score indicates a greater intensity of pain.
Time Frame: Week 12
Population: ITT; (N) = number of subjects with analyzable data at observation for pregabalin and placebo, respectively; Week 12/Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 109
scores on scale
  Burning Pain (n=108, 108) | 2.6 (0.22) | 2.9 (0.23)
  Pressing Pain (n=108, 107) | 2.7 (0.18) | 2.6 (0.19)
  Paroxysmal Pain (n=108, 108) | 1.9 (0.18) | 2.1 (0.18)
  Evoked Pain (n=108, 108) | 2.8 (0.19) | 3.2 (0.19)
  P/D (n=108, 108) | 2.7 (0.20) | 3.1 (0.20)
  Total Score (n=108, 107) | 25.7 (1.36) | 28.5 (1.40)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Burning Pain Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.216, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.2], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Pressing Pain Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.760, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = 0.1, 95% CI [-0.4 to 0.6], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.360, ANCOVA — Estimated from ANCOVA (general linear model) general linear model with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -0.2, 95% CI [-0.7 to 0.3], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Evoked Pain Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.239, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -0.3, 95% CI [-0.8 to 0.2], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; P/D Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.118, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.1], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Total Score Week 12 [LOCF]; Modelled Results; Test type: Superiority or Other; p = 0.138, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -2.8, 95% CI [-6.5 to 0.9], Standard Error of Mean 1.87

8. Secondary Outcome: Medical Outcome Study (MOS) Sleep Scale
Description: MOS: subject rated questionnaire to assess sleep quality and quantity. Consists of a 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); 7 subscales rated 1 (all the time) to 6 (none of the time): sleep disturbance, snoring, awaken short of breath (SOB) or with a headache, somnolence adequacy, and sleep quantity. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); total score range = 0 to 100; higher score indicates greater intensity of attribute.
Time Frame: Week 12
Population: ITT; (n) = number of subjects with analyzable data at observation for pregabalin and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 109
scores on scale
  Sleep disturbance (n=100, 97) | 27.1 (2.00) | 31.9 (2.05)
  Snoring score (n=98, 97) | 40.6 (2.68) | 32.9 (2.75)
  Awaken SOB or headache (n=99, 97) | 11.3 (1.95) | 15.0 (1.99)
  Sleep quantity (100, 97) | 7.0 (0.12) | 6.6 (0.12)
  Sleep adequacy (n=99, 97) | 67.5 (2.48) | 58.9 (2.51)
  Somnolence (n=99, 97) | 39.9 (1.81) | 37.8 (1.84)
  Overall sleep problems index (n=100, 97) | 28.2 (1.53) | 32.4 (1.57)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Sleep disturbance; Modelled Results; Test type: Superiority or Other; p = 0.086, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and the baseline assessment as a covariate; Mean Difference (Final Values) = -4.8, 95% CI [-10.3 to 0.7], Standard Error of Mean 2.79
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Snoring score; Modelled Results; Test type: Superiority or Other; p = 0.039, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 7.7, 95% CI [0.4 to 15.1], Standard Error of Mean 3.72
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Awaken SOB or headache; Modelled Results; Test type: Superiority or Other; p = 0.169, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI [-9.1 to 1.6], Standard Error of Mean 2.71
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Sleep quantity; Modelled Results; Test type: Superiority or Other; p = 0.030, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI [0.0 to 0.7], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Sleep adequacy; Modelled Results; Test type: Superiority or Other; p = 0.013, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 8.6, 95% CI [1.8 to 15.4], Standard Error of Mean 3.44
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Somnolence; Modelled Results; Test type: Superiority or Other; p = 0.399, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI [-2.8 to 7.1], Standard Error of Mean 2.51
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Overall sleep problems index; Modelled Results; Test type: Superiority or Other; p = 0.049, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -4.2, 95% CI [-8.4 to -0.0], Standard Error of Mean 2.13

9. Secondary Outcome: Number of Subjects With Yes or No Response for Medical Outcome Study (MOS) Sleep Scale - Optimal Sleep
Description: MOS: subject rated questionnaire to assess sleep quality and quantity. Optimal sleep component is derived from Sleep Quantity average hours of sleep each night during the past 4 weeks. Number of subjects with response = YES if sleep quantity is 7 or 8 hours per night or response = NO if sleep quantity is < 7 hours per night.
Time Frame: Week 12
Population: ITT
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 97
participants
  Optimal sleep = Yes | 51 | 42
  Optimal sleep = No | 49 | 55
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.201, Regression, Logistic — Estimated from a logistic regression model with treatment and the baseline assessment as factors; Odds Ratio (OR) = 1.5, 95% CI [0.8 to 2.9], Standard Error of Mean 0.50 — Standard error of the mean = standard error of the odds ratio

10. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - ITT Population
Description: HADS is subject rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Week 12
Population: ITT; Week 12 [LOCF]
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 108 | 108
scores on scale
  Week 12 [LOCF] Anxiety score | 5.5 (0.29) | 6.5 (0.30)
  Week 12 [LOCF] Depression score | 6.7 (0.30) | 6.5 (0.30)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 12 [LOCF] Anxiety score; Modelled Results; Test type: Superiority or Other; p = 0.015, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = -1.0, 95% CI [-1.8 to -0.2], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 12 [LOCF] Depression score; Modelled Results; Test type: Superiority or Other; p = 0.600, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = 0.2, 95% CI [-0.6 to 1.0], Standard Error of Mean 0.41

11. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Week 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 98 | 97
scores on scale | 0.5 (0.03) | 0.5 (0.03)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.566, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors and baseline score as a covariate; Mean Difference (Final Values) = 0.0, 95% CI [-0.1 to 0.1], Standard Error of Mean 0.04

12. Secondary Outcome: EQ-5D - VAS
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Week 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 99 | 97
scores on scale | 65.7 (1.78) | 62.7 (1.81)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.220, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and coutntry as factors and baseline score as a covariate; Mean Difference (Final Values) = 3.0, 95% CI [-1.8 to 7.9], Standard Error of Mean 2.47

13. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC: subject rated instrument to measure subject's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 99 | 97
scores on scale | 2.9 (0.10) | 3.1 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.144, ANCOVA — Estimated from ANCOVA (general linear model) with treament and country as factors; Mean Difference (Final Values) = -0.2, 95% CI [-0.5 to 0.1], Standard Error of Mean 0.14

14. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: CGIC: clinician rated instrument that measures change in a subject's ovall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 101 | 97
scores on scale | 2.8 (0.10) | 3.1 (0.11)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Modelled Results; Test type: Superiority or Other; p = 0.049, ANCOVA — Estimated from ANCOVA (general linear model) with treatment and country as factors; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to -0.0], Standard Error of Mean 0.14

15. Secondary Outcome: Quantitative Assessment of Neuropathic Pain (QANeP) - Sensory Threshold
Description: QANeP: assessment of sensory threshold: subject responds "yes" when monofilament stimulus is felt on area of maximum pain: 1 (lowest/softest 0.07 gram [g]) to 6 (highest 300 g) or 7 (not perceived); rated by lowest/softest filament felt when in contact with the skin. Summarized as change from baseline (mean at observation minus mean at baseline).
Time Frame: Baseline, Week 12
Population: ITT; Week 12 [LOCF].
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 106 | 107
scores on scale | 0.0 (0.89) | -0.1 (0.83)

16. Secondary Outcome: QANeP - Pain Rating Scales
Description: Subject rated pain scale: static mechanical allodynia (SMA) gentle constant mechanical pressure; dynamic mechanical allodynia (DMA) gentle stroking with foam brush; punctate hyperalgesia (PH) pinprick; cold allodynia (CA) touch with cool metal rod 13-17° celsius (C); cold hyperalgesia (CH) touch with cold metal rod 4° C; temporal summation to tactile stimuli (TSTS) repeated touching/tapping. 11-point numeric scale; range 0 (no pain) to 10 (worst possible pain). Reference area=mirror image of pain site (test area). Summarized as change from baseline (mean at observation minus mean at baseline).
Time Frame: Baseline, Week 12
Population: ITT; (n) = number of subjects with analyzable data at observation for pregabalin and placebo, respectively; Week 12 [LOCF].
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 109
scores on scale
  SMA (n=108, 107) | -0.7 (2.14) | -0.5 (1.93)
  DMA (n=108, 107) | -0.8 (1.96) | -0.6 (1.83)
  PH reference area (n=108, 107) | -0.2 (2.60) | -0.2 (2.41)
  PH test area (n=108, 107) | -0.7 (2.27) | -0.0 (2.37)
  TSTS (n=108, 106) | -1.0 (2.47) | -0.5 (2.25)
  CA (n=108, 106) | -1.1 (2.36) | -0.3 (1.95)
  CH reference area (n=107, 107) | 0.0 (2.56) | -0.2 (1.74)
  CH test area (n=107, 106) | -0.9 (2.47) | -0.9 (2.14)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 6/110 | 2/109
Other Adverse Events (participants affected / at risk) | 59/110 | 25/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=110) | Placebo (N=109)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Edema peripheral (General disorders) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=110) | Placebo (N=109)
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Oedema (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Weight increased (Investigations) | 6 | 2
Dizziness (Nervous system disorders) | 31 | 8
Headache (Nervous system disorders) | 7 | 8
Somnolence (Nervous system disorders) | 24 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.